CLINICAL TRIAL: NCT06703060
Title: Trauma-Informed HIV Prevention for Black Women in Baltimore
Brief Title: A Multi-Level Trauma-Informed Approach to Increase HIV Pre-exposure Prophylaxis Initiation Among Black Women
Acronym: MATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00018632; R01MD019178 (NIH)
Record Dates: First submitted 2024-11-07; First posted 2024-11-25 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: HIV Prevention; PrEP; Women; Intimate Partner Violence (IPV)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Peer Navigation) (Experimental): Participants randomized to this arm will receive 4 weekly group sessions and 4 one-on-one sessions with a peer navigator
  Interventions: Behavioral: Peer Navigation Group
- Control Group (Placebo Comparator): Participants randomized to this group will receive a single group session
  Interventions: Behavioral: Peer Navigation Group

INTERVENTIONS:
Behavioral: Peer Navigation Group — Participants randomized to the intervention will receive behavioral lifestyle education on topics related to biomedical HIV prevention. This will include 4 group sessions and 4 one-on-one sessions with a peer navigator.

SUMMARY:
U.S. epidemiological data indicates that Black women are a high-risk HIV disparity group, yet initiation of novel prevention strategies like pre-exposure prophylaxis (PrEP) among this group is stagnant. Socio-structural challenges like intimate partner violence and gendered racism can constrain PrEP access among Black women, but few implementation studies have mitigated these challenges to improve PrEP initiation. The proposed research aims to implement and assess the effectiveness, implementation, and sustainability of a multilevel intervention to increase PrEP initiation among Black women with and without intimate partner violence in Baltimore.

ELIGIBILITY:
Inclusion Criteria:

* self-identified Black cisgender woman;
* self-reported HIV-negative status, and
* ≥18 years.
* reports unprotected vaginal or anal sex in the past 6 months with a male sexual partner,
* have at least one substantial HIV risk factor in the past 6 months according to the 2021 Centers for Disease Control (CDC) PrEP Eligibility Guidelines (i.e., HIV-positive sexual partner, recent bacterial Sexually Transmitted Disease (STD), 2+ sex partners, history of inconsistent or no condom use, commercial sex work, and residing in high HIV prevalence area or network), and
* never taken PrEP

Exclusion Criteria:

* non-English speaking and
* currently living with HIV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender Black women (Black women who were born with female genital and also identify as women)
Enrollment: 300 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation | Post baseline up to 6 months
  Self-report of oral or injectable PrEP (Cabotegravir). Assessed from date of the most recent prescription.

SECONDARY OUTCOMES:
PrEP adherence | 2-months post-randomization, 4-months post-randomization, and 6-months post-randomization
  Biological assess of tenofovir (TFV) levels in client's urine

CONTACTS AND LOCATIONS:
Overall Officials: Tiara C. Willie, PhD, MA, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy, confidentiality, and ethical considerations. Protecting personal information is essential to comply with privacy laws (e.g., HIPAA) and the terms of informed consent. Sharing such data could breach confidentiality agreements and potentially expose sensitive information, even if anonymized. Additionally, there are concerns about data security, misuse, and the potential harm to participants, which researchers must carefully consider.